CLINICAL TRIAL: NCT06390423
Title: Passive Leg Raise and Mini-fluid Challenge Effect on Various Cardiac Output Surrogates Such as Pulse Pressure Variation (PPV), End-tidal CO2 (Carbon Dioxide), Bioreactance (Stroke Volume Index -SVI) and Velocity Time Integral on Echocardiographic Exam for Fluid Responsiveness in Patients With Moderately Severe ARDS (Acute Respiratory Distress Syndrome)
Brief Title: Passive Leg Raise and Mini-fluid Challenge Effect on Various Cardiac Output Surrogates for Fluid Responsiveness
Acronym: PHOENIX
Status: Recruiting | Type: Observational
Sponsor: CentraCare (Other)
Responsible Party: Principal Investigator, Ramakanth Pata, Principal Investigator, CentraCare
Other Study IDs: RAMPHOENIX
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Fluid Responsiveness
Keywords: Pre-load responsiveness; Passive leg raise; Mini-fluid challenge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fluid responder: Stability of vasopressor dose with maximum of 500 cc of crystalloids
  Interventions: Diagnostic Test: Passive leg raise, SVI via bioreactance, Echo based VTI
- Fluid non responder: Escalating dose of vasopressors despite 1 L of crystalloid fluid challenge

INTERVENTIONS:
Diagnostic Test: Passive leg raise, SVI via bioreactance, Echo based VTI — No interventions other than fluid challenge
  Groups: Fluid responder

SUMMARY:
In the critically ill population, fluid administration in an unstable patient is perhaps the most common intervention that is performed. Uncorrected hypovolemia with inappropriate vasopressors lead to organ hypoperfusion where as overzealous fluid administration especially in ARDS (Adult respiratory distress syndrome) can increase mortality. It has been estimated that only 50% of hemodynamically unstable critically ill patients are volume responsive, hence dynamic assessment of preload responsiveness has been proposed to better identify those individuals who would benefit from fluid bolus.

DETAILED DESCRIPTION:
Fluid responsiveness in patients with moderate to severe ARDS is crucial, as additional unnecessary fluid may be harmful. Various techniques of hemodynamic assessment exist, each with its own advantages and limitations. This study compares different techniques of preload responsiveness that include passive leg raise (PLR) and mini-fluid challenge induced changes in Pulse pressure variation (PPV), End tidal CO2, Bioreactance based Stroke volume index (SVI) and velocity time integral (VTI) on Echocardiogram.

Study protocol :

Baseline Echo with VTI will be obtained Bed side monitor will be set to display PPV and end tidal CO2 Baxter Starling system will be connected to the patient All baseline values will be recorded Tidal volume will be temporarily adjusted to 8 ml/kg , which will be reverted back to 6ml/kg after the measurements. This has proven to be a safe maneuver.

All the above hemodynamic assessments will be performed for eligible patients by measuring before and after PLR and repositioning to baseline. VTI will be estimated by bed side Echocardiogram. SVI will be estimated using the Starling system (Baxter). PPV and End tidal CO2 will be recorded from the bed side monitors.

Fluid responsiveness is presumed with a change in VTI of 10%. For these patients a mini-fluid challenge of 250 cc of crystalloids (NS, RL or Normosol) will be given over 10 min and PPV, VTI, End tidal CO2 and SVI will be recorded before and after fluid challenge. Patients with VTI change of < 10%, as non-responders, who will also be included in the analysis for assessment of reliability using the ROC curves. hemodynamic assessments and repeated fluid challenge will be considered as needed. Stability of vasopressor dose with maximum of 500 cc of crystalloid will be considered as positive fluid responder. This cohort of patients will be considered as gold standard for preload responsiveness and will be categorized based on a nominal scale. Patients who need higher vasopressor support despite 1L of crystalloid within 3 hours will be considered fluid non-responders.

Data collection:

De-identified data will be recorded. Age, BMI ( body mass index), Charleston co-morbidity index, baseline PPV, End-tidal CO2, SVI, VTI, post PLR, post fluid challenge, return to baseline, PF ratio, PEEP (positive end-expiratory pressure), SOFA (sequential organ function assessment) Score on the day of the test will be recorded.

Statistical Analysis:

Microsoft Excel will be used to record data on an institutional computer. Once the data is collected, it will be exported for statistical analysis. Jamovi will be utilized for statistical analysis. Baseline characteristics will be compared using a T-test if normative distribution or non-parametric test such as Mann Whitney U test. Reliability and accuracy will be detected using ROC curve assessment. In addition, the Youden index approach will be utilized to identify cut-offs of each of the variables and their change. (PPV, SVI,VTI and End tidal CO2). All the delta values will be compared with pearson correlation with a scatter plot and line of identity. Agreement between variables will be done using Bland-Altman analysis. If necessary, values will be transformed into Z scores. For all comparisons, a p-value of <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 - 90 years
* Diagnosis of Vasodilatory Shock with no other obvious cause of hypotension
* Diagnosis of ARDS with PF ratio < 150 , PEEP > 8
* Patients who are under paralysis or deeply sedated, on a mechanical ventilator

Exclusion Criteria:

* Patients with arrhythmias including atrial fibrillation
* Patients with chest tube, intra-abdominal hypertension or with its risk factors
* Patients with structural heart disease including pulmonary hypertension (RVSP > 45) and heart failure
* Patients on extracorporeal support such as ECMO, CRRT or MCS.
* Patients with COPD with a premorbid FEV1 < 1.5 L
* Severe atherosclerotic vascular disease

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening criteria:
  1. New onset of hypotension: MAP < 65 mm HG for > 5 min
  2. Escalation in Nor-epinephrine needs> 0.03 ug/kg/min
  3. High MAP goal Low Urine output < 0.5ml/kg/hr for > 2 hours Elevated Lactate > 4 moles/L Decreased Lactate clearance (< 40%)
  4. Bedside Echo Inc. VTI No obvious Hypovolemia No Low EF or No Pericardial effusion
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Vasopressor dose in Nor-epinephrine equivalents (NE) measured as mcg/kg/min | 3 hours after the initial passive leg raise
  We shall assess the need for vasopressor dose e.g nor-epinephrine dose. If the dose remains constant after fluid bolus until 3 hours, we shall consider them fluid resposive. If the dose requirement goes up despite fluid bolus, we shall label them fluid un-responsive

CONTACTS AND LOCATIONS:
Overall Officials: Ramakanth Pata, MD FCCP, Principal Investigator — Centracare health System
Locations (1):
- St Cloud Hospital, Saint Cloud, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monnet X, Teboul JL. Passive leg raising: five rules, not a drop of fluid! Crit Care. 2015 Jan 14;19(1):18. doi: 10.1186/s13054-014-0708-5. No abstract available. PMID 25658678
- [Background] Monnet X, Bataille A, Magalhaes E, Barrois J, Le Corre M, Gosset C, Guerin L, Richard C, Teboul JL. End-tidal carbon dioxide is better than arterial pressure for predicting volume responsiveness by the passive leg raising test. Intensive Care Med. 2013 Jan;39(1):93-100. doi: 10.1007/s00134-012-2693-y. Epub 2012 Sep 19. PMID 22990869